CLINICAL TRIAL: NCT07275359
Title: Investigating Senolytic Properties in Pulmonary Rehabilitation and Metformin in COPD Exacerbations
Acronym: INSPIRE-COPD-E
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00116416; 1K76AG095138-01 (NIH)
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD Exacerbation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: All participants will receive open-label Metformin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin (Experimental): Metformin in COPD patients without diabetes
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — All enrolled participants will receive open-label Metformin for a treatment period of 6 months.

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of Metformin and how it changes blood markers associated with aging in persons who have chronic obstructive pulmonary disease (COPD) who do not have diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* History of COPD defined by spirometry demonstrating FEV1/FVC < 70%
* 10 or more tobacco pack year history
* History of frequent exacerbations defined as: 1 severe (i.e., COPD hospitalization) or 2 moderate (i.e., outpatient treated exacerbations) in the previous 12 months

Exclusion Criteria:

* Diabetes or actively being treated with metformin
* Metformin allergy
* History of lactic acidosis not explained by acute, severe illness
* History of low vitamin B12 levels and unwilling to begin standard of care treatment for low vitamin B12 levels
* Hepatic impairment defined as history of cirrhosis or abnormal liver function tests (e.g., alanine transaminase (ALT): 7-55 units per liter (U/L), aspartate transaminase (AST): 8-48 U/L, alkaline phosphatase (ALP): 40-129 U/L, or bilirubin: 0.1-1.2 milligrams per deciliter (mg/dL))
* Renal impairment defined as eGFR < 60 mL/min/1.73m2
* Cognitive impairment
* Dementia
* Heart failure with reduced ejection fraction < 50%
* Alcohol use disorder
* Disability preventing in-person visits
* Persons with an unstable medical condition (including but not limited to unstable angina, acute heart failure exacerbation, acute neurological symptoms) or COPD exacerbation within 30 days prior to enrollment will be excluded
* Active treatment with Carbonic Anhydrase Inhibitors including but not limited to topiramate, zonisamide, acetazolamide, diclofenamide

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Determine feasibility of metformin administration in older persons with COPD without diabetes | 6 months
  Enroll and retain ≥ 30 (66%) participants through 6 months study period
Determine acceptability of metformin administration in older persons with COPD without diabetes | 6 months
  ≥70% completion of daily symptom diaries & weekly adherence logs
Determine safety of metformin administration in older persons with COPD without diabetes | 6 months
  ≥90% of the blood glucose levels, renal and hepatic function will be within normal limits*; All lactate levels will be normal
Determine tolerability of metformin administration in older persons with COPD without diabetes | 6 months
  Adverse events and Serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Mosher, MD, Principal Investigator — Duke University
Locations (1):
- Duke Asthma, Allergy, and Airway Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No